CLINICAL TRIAL: NCT01428895
Title: A Prospective Cohort Study of the Role of Surgery and/or Radiotherapy for Bone Metastases of the Femur at High Risk of Pathological Fracture
Brief Title: Femoral Bone Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OCREB 09-004
Record Dates: First submitted 2011-05-19; First posted 2011-09-05 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Cancer; Metastatic Malignant Neoplasm to Femur; Risk of Fracture
Keywords: Bone Metastases; Femoral Metastases
MeSH Terms: conditions — Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgery Alone (Active Comparator)
  Interventions: Procedure: Surgery Alone
- Surgery + Radiation Therapy (Active Comparator)
  Interventions: Other: Combined Surgery and Radiation therapy

INTERVENTIONS:
Procedure: Surgery Alone — Although we are looking at two groups, this intervention is not protocol specific but is part of the patient's standard management plan. The protocol specific part of the study is completely observational. This involves data being recorded by the attending physician during assessment and patient accounts recorded in the form of questionnaires.
  Arms: Surgery Alone
Other: Combined Surgery and Radiation therapy — Although we are looking at two groups, this intervention is not protocol specific but is part of the patient's standard management plan. The protocol specific part of the study is completely observational. This involves data being recorded by the attending physician during assessment and patient accounts recorded in the form of questionnaires.
  Arms: Surgery + Radiation Therapy

SUMMARY:
Bone is a common site of metastasis for a range of malignancies. Bone metastases have the potential to cause significant morbidity including pain, impairment of ambulation and reduced functional independence. Previous research has shown that pathological fractures are observed in 9 to 29 percent of patients with long bone metastases, and a high proportion of these require surgical intervention to relieve pain and restore function.

The goal of this study is to describe the clinical outcomes of patients with femoral metastases at high risk of pathological fracture. Patients referred for treatment of femoral metastases at high risk of fracture will be followed prospectively after undergoing with surgery (± post-operative radiotherapy), or radiotherapy alone. Patient and disease characteristics, ambulatory status and limb function will be documented before treatment. These Clinical outcomes of participants in each treatment group will be measured 6 weeks after treatment, and 3- and 6 months after enrolment, with particular reference to patient-reported outcomes relating to pain, ambulatory status, limb function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignancy other than lymphoma
* Presence of femoral metastases at high risk of pathologic fracture (Mirels' score 8 or more)
* At least 18 years of age
* Able to provide written informed consent
* Able to participate in follow-up

Exclusion Criteria:

* Surgical consultation for the purpose of obtaining a tissue/histological diagnosis only, not for treatment
* Histological diagnosis of lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2009-03; Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
To describe the ambulatory status at 3 months by intervention (surgery ± radiotherapy, and radiotherapy alone group) - Ambulatory status | 6 months
  Patient will be assessed at baseline, 6 weeks, 3 months and 6 months

SECONDARY OUTCOMES:
To describe patterns of management in patients with femoral metastases at high risk of pathological fracture - Perioperative Morbidity and Mortality for surgical patients; pain score and performance status; QOL | 6 months
  Patients will be assessed at baseline, 6 weeks, 3 months and 6 months
To describe patient and disease characteristics of major management groups (surgery ± radiotherapy, radiotherapy alone due to preference, radiotherapy alone due to co-morbid conditions) - Assessment of lower limb function | 6 months
  Patient will be assessed at baseline, 6 weeks, 3 months, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wong, MB ChB, Principal Investigator — University Health Network, Princess Margaret Hospital; Peter Ferguson, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Princess Margaret Hospital, Toronto, Ontario